CLINICAL TRIAL: NCT02072798
Title: Antibiotic Prophylaxis for Postpartum Infections Following Caesarean Section
Brief Title: Antibiotics and Gut Microbiota Among Newborn Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Copenhagen (Other); Aase and Ejnar Danielsens Foundation (Other); Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Nana Hyldig, PhD Student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s-20130117; 2012-002068-29 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-02

CONDITIONS: Surgical Wound Infection; Infection; Cesarean Section; Complications; Cesarean Section
Keywords: Randomized Controlled Trial; Caesarean Section; Surgical Site Infections; Wound Infections; Infectious Morbidity
MeSH Terms: conditions — Surgical Wound Infection; Infections; Wound Infection | interventions — Cefuroxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preoperative antibiotic (Active Comparator): iv Cefuroxime 1,5g administered 15-60 minutes before incision
  Interventions: Drug: Cefuroxime
- postoperative antibiotic (Active Comparator): iv Cefuroxime 1,5g administered after umbilical cord clamping
  Interventions: Drug: Cefuroxime

INTERVENTIONS:
Drug: Cefuroxime — iv Cefuroxime 1,5g administered 15-60 minutes before incision versus iv Cefuroxime 1,5g administered after umbilical cord clamping
  Other Names: Cefuroxime "Fresenius Kabi"

SUMMARY:
Background Women undergoing Caesarean Section (CS) have an increased risk of postpartum infections compared to women undergoing vaginal delivery. In Denmark the incidence of post-CS infections is 7-10%. The most common infections are endometritis, Urinary tract infections (UTI) and wound infections (WI).

Prophylactic antibiotics are effective in preventing postoperative infections and national guidelines recommend that antibiotics should be administered as a single dose immediately before surgical incision. CS is an exception to this pre-incision administration approach. National guidelines recommend administration of antibiotics after umbilical cord clamping to avoid exposure of the child to antibiotics before birth. Recent studies of antibiotic prophylaxis for CS suggest that prophylactic antibiotics administered before incision compared to after umbilical cord clamping may reduce post-CS infections by up to 50%. Two Cochrane reviews from 2012 criticize these types of studies for lack of data for outcomes on the baby and on late infection in the mother.

At birth, all mammals must rapidly adapt to intake of complex milk nutrients via the gut and simultaneously tolerate the invasion of billions of microbes. This requires rapid maturation of the digestive and immune functions to avoid gut disorders and infections. Full-term, breast-fed infants normally adapt well, but factors such as caesarean birth, high hygiene levels, antibiotics treatment and formula feeding may inhibit immune development both short and long term. Birth by caesarean section in high-hygiene hospital environments, and widespread use of antibiotics, are factors that reduce gut microbiota density and diversity in the newborn for some time after birth. On the other hand, high-hygiene environments and antibiotics are essential tools to combat infections, especially for the weakest newborn infants.

This pilot study will be a feasibility study to the original study, which examines the effect of change in timing of prophylactic antibiotics on the rate of post-CS infections (endometritis, UTI and WI). The pilot study focus on antibiotic and changes in the gut microbiota of newborn infants. The feasibility study will only include pregnant women in Odense with a body mass index below 30, and planned cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Women, who can read and understand Danish
* A gestational age ≥ completed 28 weeks of gestation
* Rupture of membranes and active labour (uterine contractions) is allowed.
* BMI < 30

Exclusion Criteria:

* Hypersensitivity to cefuroxime or to any other cephalosporin antibiotics
* Previous immediate and/or severe hypersensitivity reaction to penicillin or any other beta-lactam antibiotic.
* Systemic exposure to any antibiotic agent within 1 week before delivery Antibiotic indicated due to PROM, fever, group B Streptococcus or other indications at the time of caesarean section.
* Women being immunologically incompetent (e.g. HIV positive)
* Very sick newborn infants transferred to a neonatal intensive care unit and treated with antibiotics will be excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Maternal: incidence of post-CS infection (endometritis, urinary tract infections and wound infection) in each study group | Within the first 30 days after surgery
Infant: fecal microbiota at the tenth day of life | on the tenth day of life

SECONDARY OUTCOMES:
Maternal: Length of hospitalization | Within the first 30 days after Caesarean Section
Maternal: readmissions to hospital on suspicion of postpartum infection following cesarean section | Within the first 30 days after Caesarean Section
Antibiotic treatment | within the first 30 days after Caesarean Section
Infant: concentration of cefuroxime in blood samples | during the first 24 hours of life
Infant: immunological analyses in blood samples on day 3 | On the third day of life

CONTACTS AND LOCATIONS:
Overall Officials: Nana Hyldig, PhD student, Study Chair — Odense University Hospital, department of Plastic Surgery, University of Southern Denmark, Faculty of Health Sciences, institute of Clinical Research, research unit, department of Gynaecology and Obstetrics
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Kamal SS, Hyldig N, Krych L, Greisen G, Krogfelt KA, Zachariassen G, Nielsen DS. Impact of Early Exposure to Cefuroxime on the Composition of the Gut Microbiota in Infants Following Cesarean Delivery. J Pediatr. 2019 Jul;210:99-105.e2. doi: 10.1016/j.jpeds.2019.03.001. Epub 2019 Apr 30. PMID 31053348
- See also: "The NEOMUNE centre" is a research platform aiming to improve clinical care of newborn infants, particular those born with developmental problems — http://www.neomune.ku.dk